CLINICAL TRIAL: NCT07166471
Title: Global Reference Ranges - Singapore
Acronym: GRR Singapore
Status: Not yet recruiting | Type: Observational
Sponsor: Perspectum (Industry)
Collaborators: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: EC-537
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
We aim to undertake the Global Reference Range Study (GRR) to establish a set of healthy adult reference values for measures of fibroinflammation, fat and size/volumes for the liver, and other abdominal and thoracic organs to assess, compare, and if necessary, propose ethnicity specific reference ranges for these measurements.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age
* Self-reported healthy
* Willing and able to give informed consent for participation in the study
* Willing and able to undergo an MRI

Exclusion Criteria:

* History of cardiovascular disease as follows:

  * Myocardial infarction
  * Heart failure
  * Cardiomyopathy
  * Stroke
  * Hospital admission/discharge for unstable angina
  * Heart surgery
  * Unstable angina
  * Transient ischemic attack
* Presence of CVD risk factors such as hypertension, hyperlipidaemia, Type 2 diabetes, BMI > 30 kg/m2, smoker (current/ex-smoker)
* History of non-cardiac diseases related to the lungs, liver, kidneys, pancreas or spleen judged by the study investigator as therefore unsuitable to participate in the study
* The participant may not enter the study if they have any contraindication to magnetic resonance imaging (standard MRI exclusion criteria including pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia)
* Any other cause, including a significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the participant's ability to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, aged 18 years and over.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
To determine the reference values for liver fibroinflammation in healthy adults from different ethnic groups. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Pattanshetty, Study Chair — Perspectum